CLINICAL TRIAL: NCT04963829
Title: Unripe Banana Peel Powder and Lemongrass Oil in Chronic Ulcer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Adriana Rodrigues dos Anjos Mendonça, Principal Investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Banana peel
Record Dates: First submitted 2021-06-11; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Ulcer; Healing Ulcer
Keywords: Healing Ulcer; Chronic Ulcer; Musa sapientum; Lemongrass
MeSH Terms: interventions — Collagenases; Gels

STUDY DESIGN:
Intervention Model Description: Twenty-five people, regardless of gender, participated in this study. The patients were divided into 3 groups (Control 1, Control 2 and, Study Group). The Control Group 1 (CG1) consisted of seven participants who were subjected to a standardized treatment (collagenase ointment was selected for this treatment), the Control Group 2 (CG2) accounted for seven participants who used a gel made of 10% peel powder of unripe banana (M. sapientum), and the Study Group (SG) involved eleven participants who used the abovementioned gel combined with lemongrass (Cymbopogon citratus) oil at 0.1% concentration.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group (SG) (Active Comparator): Participants who used the abovementioned gel combined with lemongrass (Cymbopogon citratus) oil at 0.1% concentration.
  Interventions: Biological: gel combined with lemongrass (Cymbopogon citratus) oil at 0.1% concentration
- Control Group 1 (CG1) (Active Comparator): Participants who were subjected to a standardized treatment (collagenase ointment was selected for this treatment),
  Interventions: Biological: Collagenase ointment
- Control Group 2 (CG2) (Active Comparator): Participants who used a gel made of 10% peel powder of unripe banana (M. sapientum)
  Interventions: Biological: Gel with 10% peel powder of unripe banana

INTERVENTIONS:
Biological: gel combined with lemongrass (Cymbopogon citratus) oil at 0.1% concentration — It is a gel that was used in chronic ulcers healing
  Arms: Study Group (SG)
Biological: Collagenase ointment — Participants who were subjected to a standardized treatment (collagenase ointment)
  Arms: Control Group 1 (CG1)
Biological: Gel with 10% peel powder of unripe banana — Participants who used a gel made of 10% peel powder of unripe banana (M. sapientum),
  Arms: Control Group 2 (CG2)

SUMMARY:
To evaluate the activity of a gel composed of 10% peel powder of unripe banana (Musa sapientum) combined with lemongrass (Cymbopogon citratus) oil, at 0.1% concentration, in patients with chronic ulcers.

DETAILED DESCRIPTION:
Purpose: To evaluate the activity of a gel composed of 10% peel powder of unripe banana (Musa sapientum) combined with lemongrass (Cymbopogon citratus) oil, at 0.1% concentration, in patients with chronic ulcers. Methods: This is a clinical, individual, analytical, interventional, longitudinal, prospective, controlled study with convenience sampling. Three groups will be used, as follows: control group 1 (CG1) with 7 participants will be treated with collagenase, control group 2 (CG2) with 7 participants will be treated with a gel composed of 10% unripe banana peel powder, and study group (SG) with 11 patients will be treated with the abovementioned gel combined with lemongrass oil at 0.1% concentration. The ulcer areas will be analyzed once a week for 4 weeks. Afterward, wound areas will be measured and the obtained data will be subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* presence of chronic ulcers,
* 18 years of age and older

Exclusion Criteria:

* Patients who had any type of allergic reaction to the study products during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Delimitation of the wound area | 3 month
  To delimit the wound area, plastic and a fine-tipped pen will be used to outline the edge of the wound.

SECONDARY OUTCOMES:
Digitalizing drawing wounds measurements | 3 months
  All collected measurements (drawings) were scanned and saved in JPEG format and the areas were calculated using the ImageJ® software13.
  The ImageJ® was set to measure the area in centimeters, with a pixel of 118.67, establishing a fixed value. The areas were calculated individually in the software and the values were saved in an Excel spreadsheet.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R dos Anjos Mendonça, PhD, Principal Investigator — Vale do Sapucaí University
Locations (1):
- Vale do Sapucaí University, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No